CLINICAL TRIAL: NCT05066945
Title: Application of Circulating Tumor (ctDNA) in the Evaluation of Curative Effect and Prognosis of Small Cell Lung Cancer (SCLC) Patients
Brief Title: Application of ctDNA in the Evaluation of Curative Effect and Prognosis of SCLC Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, dengpengbo, Attending physician, Xiangya Hospital of Central South University
Other Study IDs: 202103748
Record Dates: First submitted 2021-08-19; First posted 2021-10-04 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-09

CONDITIONS: Small Cell Lung Cancer Extensive Stage
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observation — observe the association of ctDNA with efficacy of treatment

SUMMARY:
The purpose of this study is to evaluate the application value of circulating tumor DNA(ctDNA) with efficacy evaluation and prognostic assessment in patients with unresectable SCLC, who were receiving radiotherapy and chemotherapy treatment.

DETAILED DESCRIPTION:
1. According to each point in time of ctDNA, to analyze the dynamic changes of tumor burden and clonal subtypes which to evaluate the application value of ctDNA in curative efficacy evaluation.
2. Compare the two time points before and after radiotherapy and chemotherapy treatment of the cell free DNA (cfDNA) concentration and tumor burden, analysis the correlation between the changes and prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent；
* Newly diagnosed and histological or cytological confirmed extensive stage small cell lung cancer;
* All indicators has confirmed and allow to receive radiotherapy and chemotherapy;
* Follow-up can be carried out and the peripheral blood samples can be collected;
* Cooperate with the provision of clinical pathological data required by the research.

Exclusion Criteria:

* Patients have other primary cancers;
* Patients unable to cooperate with the study for follow-up according to the determined clinical follow-up cycle;
* Unable to accept the judgment of curative effect evaluation by the designated methods such as CT.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: treatment extensive stage small cell lung cancer patients
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
ctDNA mutation profile at baseline | before treatment ctDNA mutation analysis and clonal analysis (each cycle is 3 weeks)
  ctDNA mutation will be detected, PyClone based clonal analysis will be performed to analyze the clonal dominance
the evolution of ctDNA mutation profile during treatment | After the first cycle of first line treatment upon physicians' request, ctDNA mutation analysis and clonal analysis (each cycle is 3 weeks)
  ctDNA mutation will be detected, PyClone based clonal analysis will be performed to analyze the clonal dominance
the evolution of ctDNA mutation profile during treatment | After finished the first line treatment, ctDNA mutation analysis and clonal analysis (each cycle is 3 weeks)
  ctDNA mutation will be detected, PyClone based clonal analysis will be performed to analyze the clonal dominance

SECONDARY OUTCOMES:
PFS | From the first line treatment to the time of disease progression (through study completion, an average of 5 months)
  Progression free of survival

IPD SHARING:
Plan to Share IPD: Yes
all IPD data for publication
Supporting Information: Study Protocol
Time Frame: IPD will be shared when the clinical trail is completed.

REFERENCES:
- [Background] Mohan S, Foy V, Ayub M, Leong HS, Schofield P, Sahoo S, Descamps T, Kilerci B, Smith NK, Carter M, Priest L, Zhou C, Carr TH, Miller C, Faivre-Finn C, Blackhall F, Rothwell DG, Dive C, Brady G. Profiling of Circulating Free DNA Using Targeted and Genome-wide Sequencing in Patients with SCLC. J Thorac Oncol. 2020 Feb;15(2):216-230. doi: 10.1016/j.jtho.2019.10.007. Epub 2019 Oct 16. PMID 31629061
- [Background] Nong J, Gong Y, Guan Y, Yi X, Yi Y, Chang L, Yang L, Lv J, Guo Z, Jia H, Chu Y, Liu T, Chen M, Byers L, Roarty E, Lam VK, Papadimitrakopoulou VA, Wistuba I, Heymach JV, Glisson B, Liao Z, Lee JJ, Futreal PA, Zhang S, Xia X, Zhang J, Wang J. Circulating tumor DNA analysis depicts subclonal architecture and genomic evolution of small cell lung cancer. Nat Commun. 2018 Aug 6;9(1):3114. doi: 10.1038/s41467-018-05327-w. PMID 30082701